CLINICAL TRIAL: NCT04304586
Title: Evaluating the Correlation Between the Results of the Allergy Work-up for Different Allergens of the Anacardiaceae Family
Brief Title: Clinical Cross Reactions Between Anacardiaceae
Acronym: Cross-Anacards
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0151
Record Dates: First submitted 2020-03-09; First posted 2020-03-11 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Suspected Allergy to Anacardiaceae
Keywords: Food allergy; Skin tests; Food challenge; Cashew; Pistachio
MeSH Terms: conditions — Food Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The prevalence of food allergies has increased in recent decades, ranging from 1 to 3% of the general population. According to international literature and French national surveys, nuts today represent a group of allergens often associated with severe allergic reactions. They are responsible for 18 to 40% of deaths from food-related anaphylaxis.

Among all nuts, the prevalence of anacardiac allergies (mainly cashew and pistachio) continues to increase and has become a growing public health problem. Today, global production is estimated at 4.9 million tonnes of cashews and 1.1 million tonnes of pistachios. The resulting increased exposure may explain the increased prevalence of allergic reactions reported to these fruits. In addition, anaphylactic reactions to anacardiaceae are reported to be even more severe than those occurring in subjects allergic to peanuts.

Cashews and pistachios are known to exhibit immunological cross-reactions with one another. In fact, they have a strong sequential homology between their storage allergens Ana o 1 / Pis v 3 (7S vicilin, 78% homology); Ana o 2 / Pis v 2 (legume 11S, 80% homology) and Ana o 3 / Pis v 1 (albumin 2S, 70% homology). For this reason, some authors talk about the cashew / pistachio syndrome and associate the two allergenic sources by considering them as one, in clinical practice.

The diagnosis of allergy to nuts, and therefore to anacardiaceae, is based on a compatible clinical history, the presence of specific IgE (demonstrated by positivity to realistic skin tests and serum IgE assay), and positivity on the oral food challenge test.

In clinical practice, taking into account the cashew / pistachio syndrome, when the allergy work-up for cashew is negative, allergists tend to advise to reintroduce pistachio at home, considering the two allergens as sufficiently homologous to authorize such a practice. In this context, the investigators decided to check whether this practice, which is based mainly on in vitro homologies, is risk-free, based on the clinical experience of our center.

ELIGIBILITY:
Inclusion criteria:

* Patient evaluated at the Allergy Unit of the University Hospital of Montpellier (France)
* Suspicion of food allergy to Anacardiaceae
* Allergy work-up for cashew and pistachio including at least skin tests, and possible specific IgE and food challenge

Exclusion criteria:

- Patients included in other trials that don't allow them to be included in the present one

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients consulting at the Allergy Unit of the University Hospital of Montpellier (France) for a suspected food allergy to Anacardiaceae
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2006-01-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
PPV and NPV | 1 day
  PPV and NPV of the results of skin tests and food challenge to either cashew or pistachio to predict a concordant result for pistachio or cashew, respectively

SECONDARY OUTCOMES:
Relative risk | 1 day
  Finding risk factors predictive of discrepancies between the results of the allergy work-up for cashew and pistachio

CONTACTS AND LOCATIONS:
Overall Officials: Davide CAIMMI, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC